CLINICAL TRIAL: NCT03576742
Title: Register für Schwere Immunzytopenien - Severe Immune Cytopenia Registry (SIC-Reg.Org)
Brief Title: Severe Immune Cytopenia Registry Www.Sic-reg.Org
Acronym: sic-reg
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 30-155 ex 17/18
Record Dates: First submitted 2018-06-08; First posted 2018-07-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Immune Thrombocytopenia; Autoimmune Hemolytic Anemia; Evans Syndrome; Primary Immunodeficiency
Keywords: pancytopenia; aplastic anemia; myelodysplastic syndrome; primary immunodeficiency; immune dysregulation; autoimmune cytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Evans Syndrome; Primary Immunodeficiency Diseases; Pancytopenia; Anemia, Aplastic; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — stool, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: all who fulfil inclusion criteria and consent to participation; potential biomarkers will be documented
  Interventions: Diagnostic Test: potential biomarkers

INTERVENTIONS:
Diagnostic Test: potential biomarkers — facs analysis, microbiome analysis

SUMMARY:
Prospective registry study for children and young adults with severe immune cytopenias (persisting/chronic immune thrombocytopenia, autoimmune hemolytic anemia, and Evans syndrome) to improve the management, facilitate the differential diagnostic work-up, and document the clinical course under various treatments.

Time points: at inclusion, after 6 months, after 12 months, then yearly up to 4 years after inclusion.

No intervention, mere observation and documentation. Guided pre-inclusion (differential) diagnostic work-up.

DETAILED DESCRIPTION:
The study aims to improve the management and care of patients with severe immune cytopenias, to identify underlying causes of severe immune cytopenias and to develop a strategy for early treatment stratification based on a standardized diagnostic algorithm, potentially supported by biomarker analyses and (off study) genetic analyses, where clinically indicated.

Primary Goal:

Rapid detection of underlying causes of severe immune cytopenias with the aid of a structured diagnostic approach and access to a clinical care network of the participating centers, allowing early treatment stratification

Secondary Goals:

* Collection of data about epidemiology of rare diseases
* Systemic documentation of response rates to various treatments
* Identification of biomarkers and modifiers of immune tolerance
* Collection of data about the usage of novel/experimental therapeutic agents
* Documentation of physician-reported outcome measures/performance scores
* Consultation of the caring physicians through a regular SIC-Reg board

There will be no additional venous punctures or investigational time points. At clinical visits around planned study time points, additional blood parameters and stool specimen will be obtained. The current clinical management follows international guidelines, which are summarized in the study documents but do not represent part of the study (no diagnostic or therapeutic investigational arm).

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune hemolytic anemia (AIHA)
* Evans syndrome (ES)
* Persistent or chronic immune thrombocytopenia (ITP; >6 months after first manifestation)

Exclusion Criteria:

* (history of) malignancies
* (history of) hematopoietic stem cell transplantation

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: consecutive registration of pediatric, adolescent, and young adult patients with severe immune cytopenia who consent
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
underlying disease that causes or is associated with severe immune cytopenia | 0-4 years
  identify the underlying condition or other disease, e.g., primary immunodeficiency or bone marrow failure syndrome by diagnostic procedures according to a standardized algorithm

SECONDARY OUTCOMES:
Clinical course | 0-4 years
  Documentation of physician-reported clinical symptoms including outcome measures/performance scores
Biomarkers - Blood | 0-4 years
  Identification of novel biomarkers by flow cytometry of leukocytes
Biomarkers - Stool | 0-4 years
  Identification of potential modifiers of immune tolerance by studying the intestinal microbiome
Routine laboratory parameters | 0-4 years
  documentation of laboratory parameters that are routinely assessed for immune cytopenia
Number of participants with the diagnosis of severe immune cytopenia per participating centre and per year | 0-4 years
  epidemiological data acquisition, participants included according to the inclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Seidel, Principal Investigator — Medical University of Graz
Locations (1):
- Pediatric Hematology-Oncology Outpatient Clinic, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided